CLINICAL TRIAL: NCT00230269
Title: The Role of FDG PET in Radiation Treatment Planning for Head and Neck Cancers
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Other Study IDs: ENT0005; ENT0005; NCT00230269
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: PET-CT

SUMMARY:
In patients with cancer of the head and neck and rectum, knowing the exact location of the tumor is important for designing the radiation field to ensure delivery of high dose of radiation to the tumor while sparing surrounding normal tissues. A new medical imaging method which is a combination of positron emission tomography (PET) and computed tomography (CT) scan, has shown promise in helping the radiation oncologist in defining the exact location and extent of the tumor in certain cancers such as lung cancers. Therefore the purpose of this study is to determine if these imaging methods can be used in combination with the standard radiation treatment planning procedure to improve the accuracy to targeting your tumor with radiation. In addition the PET-CT scan, similar to the PET scan alone with better resolution, can be used to determine whether the tumor has spread to any part of the body outside of the head and neck sites.

ELIGIBILITY:
Inclusion Criteria:Patients who are scheduled to receive radiation therapy for head and neck cancer at Stanford.

Exclusion Criteria:Non-Stanford patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled to receive radiation therapy for head and neck cancer at Stanford.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2003-05; Primary Completion 2006-06 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Thu Le, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States